CLINICAL TRIAL: NCT00596986
Title: Impact of Therapeutical Strategies on Emotional Processing in Depression: Neurofunctional and Clinical Issues in the Context of Affective Bias
Brief Title: Getting Biased Treatment Study: How Psychotherapy and Antidepressants Change Brain Activity in Chronic Depression
Acronym: GETTY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Dr. med. Michael Colla, Dept. of Psychiatry, Campus Benjamin Franklin, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EUK-B2.1; EUK-B2
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Depression
Keywords: Depression; Duloxetine; Psychotherapy; Magnetic Resonance Imaging
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride

ARMS (2):
- AD (Active Comparator): Antidepressant Duloxetine
  Interventions: Drug: Duloxetine
- PT (Active Comparator): Psychotherapy (CBASP) - Cognitive Behavioural Analysis System of Psychotherapy
  Interventions: Behavioral: Cognitive Behavioural Analysis System of Psychotherapy

INTERVENTIONS:
Drug: Duloxetine — Duloxetine 30mg up to 120mg per day.
  Arms: AD
Behavioral: Cognitive Behavioural Analysis System of Psychotherapy — Cognitive Behavioural Analysis System of Psychotherapy (CBASP): 20 sessions of psychotherapy, beginning with twice weekly, then weekly sessions.
  Arms: PT

SUMMARY:
The purpose of this study is to determine how psychotherapy and pharmacotherapy respectively change brain activity in patients suffering from chronic depression.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Depression (Double Depression, Chronic MDE, MDE with incomplete remission)
* HAMD-24>20

Exclusion Criteria:

* Concurrent Psychotherapy or Psychopharmacotherapy
* Previous Non-Response to Duloxetine
* Non-Response to three Antidepressants of two different groups given at adequate doses or Non-Response to two empirically tested forms of Psychotherapy in the current Depressive Episode
* Serious Psychiatric comorbidity
* Serious Neurologic comorbidity
* Contraindications to Duloxetine
* Contraindications to fMRI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Neuroimaging Data (fMRI) | Before and After Therapy

SECONDARY OUTCOMES:
HAMD | Weekly
Salivary Cortisol | Before and After Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Heuser, Prof. Dr. med. Dipl. Psych., Study Chair — Dept. of Psychiatry, Campus Benjamin Franklin, Charité Berlin, Germany; Michael Colla, Dr. med., Principal Investigator — Department of Psychiatry, Campus Benjamin Franklin, Charité Berlin, Germany
Locations (1):
- Charité Universitätsmedizin, Berlin, State of Berlin, Germany